CLINICAL TRIAL: NCT04781868
Title: Multi-Nutrient Supplement for Radio-Protection
Acronym: MNSRP
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13032
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Oxidative Stress; DNA Damage, Radiation Induced; Radiation Exposure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-nutrient supplement (Experimental)
  Interventions: Drug: Multi-nutrient supplement
- Placebo supplement (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Multi-nutrient supplement — Multi-nutrient supplement containing a combination of vitamins, minerals and antioxidants
  Arms: Multi-nutrient supplement
Drug: Placebo — Placebo
  Arms: Placebo supplement

SUMMARY:
Exposure to radiation, such as during routine CTs, bone scans, or X-rays, causes oxidative stress which can damage the DNA (your genetic material) within your white blood cells. While the amount of DNA damage that may occur from one scan is not harmful to your overall health, there could be concerning damage in patients who are constantly exposed to this radiation. Currently, there is no way to prevent DNA damage during a medical scan. One potential way to fight the oxidative stress caused by radiation is to take an antioxidant before a scan. The purpose of this study is to see if a combination of antioxidants can protect someone from the damage that radiation causes to the DNA of their white blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 76 years.
* Scheduled for bone scan procedure at the Juravinski Hospital.

Exclusion Criteria:

* History of smoking within six months prior to study enrollment.
* Known hypersensitivity reactions to any of the ingredients in the MNSRP.
* Chemotherapy or radiation therapy within six months prior or one month following study enrollment.
* Individuals currently taking vitamin or mineral supplements that contain antioxidants will be considered on a case-by-case basis but will be asked to refrain from intake for at least two weeks prior to partaking in this study.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of gamma-H2Ax foci per PBMC nucleus | Three hours following radiation exposure
  Number of gamma-H2Ax foci per PBMC nucleus three hours following radiation exposure

SECONDARY OUTCOMES:
Amount of amplifiable mtDNA in PBMC's | Three hours following radiation exposure
  Amount of amplifiable mtDNA in PBMC's three hours following radiation exposure
Abundance of mtDNA deletions in PBMC's | Three hours following radiation exposure
  Abundance of mtDNA deletions in PBMC's three hours following radiation exposure
Abundance of phosphorus-ATM in PBMC's | Three hours following radiation exposure
  Abundance of phosphorus-ATM in PMBC's three hours following radiation exposure

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol